CLINICAL TRIAL: NCT02309619
Title: Lifting of Gastric Tube Through Trans-substernal Versus Trans-esophageal Bed Path in Minimally Invasive Esophagectomy: a Single-Center Randomized Controlled Trial
Brief Title: Lifting of Gastric Tube Through Trans-substernal Versus Trans-esophageal Bed Path in MIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Kun Li, MD, Kun Li, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kli
Record Dates: First submitted 2014-11-23; First posted 2014-12-05 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Esophageal Neoplasms; Esophagectomy
Keywords: esophageal cancer; esophagectomy; quality of life
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trans-substernal group (Experimental): Patients who undergo esophagectomy with the gastric tube lifting to the neck through trans-substernal path.
  Interventions: Procedure: lifting of the gastric tube to the neck for gastro-esophageal anastomosis through trans-substernal or trans-esophageal bed path.
- trans-esophageal bed group (Experimental): Patients who undergo esophagectomy with the gastric tube lifting to the neck through trans-esophageal bed path.
  Interventions: Procedure: lifting of the gastric tube to the neck for gastro-esophageal anastomosis through trans-substernal or trans-esophageal bed path.

INTERVENTIONS:
Procedure: lifting of the gastric tube to the neck for gastro-esophageal anastomosis through trans-substernal or trans-esophageal bed path. — Patients with esophageal cancer (EC) will undergo minimally invasive esophagectomy and be classified into two groups according to the last step of the procedure. The gastric tube will be lifted to the neck for gastro-esophageal anastomosis through trans-substernal path in the trans-substernal group, and through trans-esophageal bed path in the trans-esophageal bed group.

SUMMARY:
Esophageal cancer (EC) is the eighth most common cancer and the sixth leading cause of cancer deaths worldwide. Minimally invasive esophagectomy (MIE) is regarded as a safe and effective management for resectable EC. Gastric tube is considered to be an ideal substitute for the resected esophagus and can be lifted to the neck for anastomosis through two different paths - Trans-substernal and trans-esophageal bed routes. However, the differences of operative outcomes between the two paths have not been systematically described. In this study, clinical outcomes including intra- and post-operative status, morbidity and complications, nutrition status, as well as quality of life after surgery will be evaluated, and differences between the trans-substernal and trans-esophageal bed groups will be compared. The study might help to individualization treatment for EC.

DETAILED DESCRIPTION:
1. Patients with esophageal cancer (EC) will be histologically proved by endoscopic biopsy, and staged by thoracicoabdominal computed tomography (CT), endoluminal ultrasonography and positron emission tomography (PET) before surgery. The other crucial test including barium meal, pulmonary function tests, arterial blood gas analysis, cardiac ultrasonography, electrocardiogram and treadmill test, as well as blood biochemistry examinations will also be accomplished preoperatively.
2. Patients who meet clinical criteria will be asked to sign a consent form, and divided randomly into two groups - trans-substernal group and trans-esophageal bed group. Patients in both groups will undergo a minimally invasive esophagectomy which consist of 4 steps: (1) thoracoscopic esophageal mobilization followed by mediastinal lymphadenectomy; (2) laparoscopic gastric mobilization followed by abdominal lymphadenectomy and gastric tube construction; (3) cervical esophageal mobilization and transection; (4) lifting of the gastric tube to the neck for gastro-esophageal anastomosis through trans-substernal or trans-esophageal bed path. The operative procedure of the two groups is similar except step 4.
3. Patients in both groups will be followed-up regularly. Intra- and post-operative status, morbidity and complications, nutrition status, as well as quality of life after surgery will be evaluated, and differences between the trans-substernal and trans-esophageal bed groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma, adenocarcinoma or undifferentiated carcinoma of the intrathoracic esophagus.
* Surgical resectable (T1-4a, N0-3, M0).
* Age ≥ 18 and ≤ 75 years.
* European Clinical Oncology Group (ECOG) performance status 0,1 or 2.
* Written informed consent obtain

Exclusion Criteria:

* Carcinoma of the cervical esophagus.
* Carcinoma of the gastro-esophageal junction (GEJ).
* Prior thoracic surgery or trauma on the right hemithorax, or previous diseases which may lead to right pleural adhesion (these patients will undergo open surgery instead of minimally invasive esophagectomy).
* Dysfunction of cardiorespiratory system or other surgical contraindications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Composite intra-operative features. | During the operation (an expected average of 5 hours).
  The composite intra-operative features of patients in trans-substernal and trans-esophageal bed paths will be evaluated and the results will be compared. These intra-operative features will be composed of duration of operation (min), estimated blood loss (ml), mean arterial pressure (mmHg), central venous pressure (cmH2O), heart rate (beat/min), stroke volume variation (%), cardiac output (L/min), cardiac index (L/m2min) and stroke volume index (ml/m2).
Composite post-operative features. | From the day of operation to hospital discharge (an expected average of 2 weeks).
  The composite post-operative features of patients in trans-substernal and trans-esophageal bed paths will be evaluated and the results will be compared. These post-operative features will be composed of duration of ventilation (hours), duration of chest tube drainage (days), duration of stomach tube drainage (days), duration of duodenal feeding (days), duration of parenteral nutrition (days), duration of fasting (days), duration of systemic inflammatory response syndrome (days), duration of ICU stay (days), duration of postoperative hospital stay (days), gastric fluid drainage (ml), number of transfused patients (%) and expense (thousand yuan).
Mortality and complications. | From the day of operation to hospital discharge (an expected average of 2 weeks).
  Mortality and complications of patients with the gastric tube lifted through trans-substernal and trans-esophageal bed paths will be evaluated and the results will be compared. These parameters will be composed of in-hospital/30-day mortality, respiratory failure/adult respiratory distress syndrome (ARDS)/reintubation, chylothorax, pleural infection, hemorrhage requiring reoperation, membranous trachea injury, deep venous thrombosis/pulmonary embolus, diaphragmatic hernia, arrhythmia, pneumonia, cervical anastomotic leak/stricture, vocal cord palsy, cervical anastomotic stricture, delayed gastric emptying and wound infection.

SECONDARY OUTCOMES:
Composite nutrition status. | Every 3 months until the 1st year after operation (follow-up for a year after surgery).
  Patients with the gastric tube lifted through trans-substernal and trans-esophageal bed paths will be followed-up regularly every 3 months during the first year after surgery. The composite nutrition status of the patients in both groups will be evaluated and the results will be compared. These nutrition status will be composed of weight change (kg), body mass index (kg/m2), body fat (%), red blood cell (10^12/L), hematocrits (%), hemoglobin (g/L), serum albumin (g/L) and serum prealbumin (g/L).
Quality of life. | Every 3 months until the 1st year after operation (follow-up for a year after surgery).
  Patients with the gastric tube lifted through trans-substernal and trans-esophageal bed paths will be followed-up regularly every 3 months during the first year after surgery. Quality of life (QOL) of the patients will be assessed using a composite cancer-specific core questionnaire, the quality of life questionnaire (QLQ)-C30 (version 3.0, in Chinese) and the esophageal module QLQ-Oesophageal(OES)18 (in Chinese) both developed by the European Organization for Research and Treatment of Cancer (EORTC), and the results will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Li, MD, Study Chair — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China